CLINICAL TRIAL: NCT06759987
Title: Construction and Application of a Self-Care Behavior Intervention Scheme for Chronic Heart Failure Patients Based on Interaction Model of Client Health Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhi-fen Feng (Other)
Responsible Party: Sponsor-Investigator, Zhi-fen Feng, associate professor, Henan University
Organization: Henan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUSOM2023-441
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Chronic Heart Failure; Self-care; Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): The control group received routine care.
- intervention group (Experimental): The intervention group received the self-care behavior intervention program based on the interaction model of health behavior.
  Interventions: Behavioral: self-care behavior intervention

INTERVENTIONS:
Behavioral: self-care behavior intervention — The intervention group received the self-care behavior intervention program based on the interaction model of health behavior
  Arms: intervention group

SUMMARY:
The purpose of this study, which will last for 3 months, is to investigate the effect of the intervention based on the interaction model of health behavior on patients' disease perception, heart failure self-care level, quality of life and service satisfaction. If you have any questions or difficulties, you can withdraw from this study at any time, which will not affect your treatment and care; The purpose of this study is to improve your level of self-care, prevent your readmission to the hospital, and do not harm your physical and mental health, nor negatively affect the patient's relationship with care; Your participation in the study and the personal data in the study are confidential, and any public report on the results of this study will not disclose your personal identity.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CHF according to the New York Heart Association (NYHA) functional classification of II-III.
* Age ≥ 18 years, stable condition, clear consciousness, normal language and written expression abilities, no communication barriers, able to understand and accurately complete questionnaires.
* Informed consent and voluntary participation.

Exclusion Criteria:

* -Patients with complications such as renal or hepatic insufficiency, a history of mental disorders, or currently experiencing mental disorders, or critically ill.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Chinese Version of the Self-Care of Heart Failure Index (SCHFI) | Baseline, one month and three months

SECONDARY OUTCOMES:
Brief Illness Perception Questionnaire (BIPQ) | Baseline, one month and three months
Minnesota Living with Heart Failure Quality of Life Questionnaire (MLHFQ) | Baseline, one month and three months

OTHER OUTCOMES:
Unplanned Readmission | one month and three months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nursing and Health, School of Nursing and Health,Henan University, Kaifeng, Henan, China

IPD SHARING:
Plan to Share IPD: No